CLINICAL TRIAL: NCT04817540
Title: Phase II Trial of Anti-HER2 Treatment in HER2-enriched Early Breast Cancer Identified by PAM50 (HER2E-PAM, PAMILIA Study)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Joon Jeong, Professor, Gangnam Severance Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3-2021-0026
Record Dates: First submitted 2021-03-25; First posted 2021-03-26 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: HER2 Enriched Subtype Breast Cancer, Herzuma, PAM50 Study

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, Herzuma arm (Experimental)
  Interventions: Drug: Herzuma

INTERVENTIONS:
Drug: Herzuma — 8mg/kg IVF loading dose at first cycle -> 6mg/kg IVF at 2,3,4th cycle of each 21 day cycle

SUMMARY:
In this study, we prospectively analyzed molecular subtyping through the PAM 50 test in HER2-negative (IHC1+ or 2+ (FISH/SISH-)) breast cancer patients. A phase 2 single arm study was designed to determine whether the addition of HER2-targeted treatment with treatment increases the pathologic remission rate.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically and cytologically documented unsectable/metastatic breast cancer that :

   A. has confirmed HER2 negative expression regardless hormone receptor status
   * definition of HER2 negative breast cancer i) HER2 IHC 1+ without ISH or ii) HER2 IHC 2+ and ISH negative (average HER2 gene copy number <4 signals/cell in single probe ISH or HER2/CEP17 ratio <2.0 & average HER2 gene copy number <4 signals cell in dual-probe ISH)
2. No prior treatment of stage II-III breast cancer

   * HR+ & HER2- breast cancer : cT1-4N1-3
   * HR- & HER2- breast cancer : cT1N1-3 or cT2-4N0-3
3. No systemic metastasis confirmed by pathological or radiological evaluation
4. Patients over 19 years
5. Confirmed to HER2-enriched subtype by PAM50 study
6. Available FFPE 15-20 slides for evaluating PAM50 study
7. ECOG 0-1
8. Adequate bone marrow functions i) Hemoglobin≥ 9g/dL ii) ANC ≥1,500/mm3 iii) Platelet ≥100,000/mm3
9. Adequate renal functions i) creatinine : ≤ 1.5 x UNL or ii) creatinine clearance (Ccr) ≥ 50 ml/min by Cockroft formula
10. Adequate liver functions i) Bilirubine : ≤ 1.5 x UNL ii) AST/ALT : ≤ 2.5 x UNL
11. Adequate cardiac functions

    * LVEF ≥50% (with MUGA scan or TTE)
12. Females of childbearing potential must have a negative serum or urine pregnancy test within 72 hours prior to first dose of study treatment.

Exclusion Criteria:

* 1) History of previous treatments of ipsilateral or contralateral invasive breast cancer 2) Confirmation of systemic distant metastasis of breast cancer 3) History of other malignancy within the last 5 years, except curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, less than 2cm of thyroid cancer (papillary, follicular, medullary).

  4) inflammatory breast cancer (cT4d) 5) bilateral breast cancer(except, multifocal or multicentric breast cancer) 6) occult breast cancer 7) History of positivity for hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus (HIV) 8) Woman of childbearing potential who is not consenting to use highly effective methods of birth control (eg, true abstinence [periodic abstinence (eg calendar ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception], sterilization, or other non-hormonal forms of contraception) during treatment 9) Uncontrolled infections and other serious diseases or medical conditions 10) Uncontrolled hyeprtension or clinically active cardiovascular disease: for example, cerebrovascular accident or transient isschemic attack, unstable angina, myocaridal infarction within 6 months prior to enrolment. Have symptomatic congestive heart failure (CHF; New York Heart Association II-IV) or symptomatic or poorly controlled cardiac arrhythmia.

  11) Have any condition (eg, psychological, geographical, or medical) that does not permit compliance with the study and follow-up procedures or suggest that the patient is, in the investigator's opinion, not an appropriate candidate for the study 12) Patients who are hypesenstivie reaction to experimental drugs (doxorubicin, cyclophosphamide, paclitaxel, docetaxel, herzuma) 13) Peripheral neuropathy CTCAE v4.03 ≥ grade 2

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-03-30 (Estimated); Study Completion 2027-03-30 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate (%, ypT0/isN0) | 12 weeks
  TPathologic Complete Response (pCR) rate, assessed as no evidence of invasive disease in excised surgical specimens of breast and/or axilla(ypT0/isYpN0), in participants who received at least 1 cycle of herzuma and taxane in HER2-enriched subtype breast cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Gangnam Severance Hospital, Seoul, South Korea